CLINICAL TRIAL: NCT01153165
Title: Pilot Study of Treatment of Depression in Refractory Asthma
Brief Title: Study of Treatment of Depression in Refractory Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liam Heaney (Other)
Collaborators: Asthma UK (Other)
Responsible Party: Sponsor-Investigator, Liam Heaney, Consultant Physician, Belfast Health and Social Care Trust
Organization: Belfast Health and Social Care Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10015LH-OPMS
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: Refractory; Asthma; Depression
MeSH Terms: conditions — Asthma; Depression | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citalopram (Experimental): Participants will be commenced on Citalopram 20mgs daily
  Interventions: Drug: Citalopram
- Control (Placebo Comparator): Control group - will receive a matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram — Participants will be commenced on Citalopram 20mgs daily. At week 4 participants will be assessed for response to treatment . If no response, dose of Citalopram will be increased to 40mgs for the remaining 8 weeks of the study. Patients who respond will remain on 20mgs for remaining 8 weeks.
  Arms: Citalopram
Drug: Placebo — Participants in the control group will receive a matched placebo. At week 4 participants will be assessed for response to treatment. If no response, dose of placebo will be increased to 40mgs for the remaining 8 weeks of the study. Patients who respond will remain on 20mgs for remaining 8 weeks.
  Arms: Control

SUMMARY:
Purpose and design: The relationship between psychological morbidity and asthma has been previously recognised, however there is little evidence regarding the link between poor mental health and asthma control in people with severe asthma. If evidence was available showing that identifying and treating depression, resulted in meaningful improvements in people's asthma symptoms, this would be helpful in changing doctors' approach to people with severe asthma, ensuring that both physical and mental wellbeing were considered.

This study will be a double blind randomised placebo controlled pilot study which aims to identify; if treating depression in patients with well characterised refractory asthma improves depression and asthma control. Forty patients who meet the inclusion criteria will be randomised to either a placebo or anti-depressant medication group, neither the participant nor the researcher will be aware of which medication they are given. Patients recruited will have severe asthma; will be identified as having depression using two validated questionnaires and will agree to take part and to take anti-depressant medication. Patients with poor adherence to medication, other respiratory conditions and who have had anti-depressant medication in previous the 6 months will be excluded. Outcome measures such as depression questionnaires, quality of life questionnaire, lung function, measures of airways inflammation and reduction in dose of oral steroids will be used to determine the effect of anti-depressant medication on depression and asthma control. The treatment period will be 12 weeks with outcomes assessed in the first and final week of treatment. The investigators hope to find out if the study protocol we have devised is feasible for a larger multi-Centre clinical trial and demonstrate some evidence that treating depression in subjects with well characterised refractory asthma will improve depression and asthma symptom control (this will be used to estimate the size of a larger clinical trial).

Recruitment: Participants will be identified and approached by a member of their usual healthcare team and invited to participate. Participants will be given time to consider whether they wish to take part and will assured that their care will be unaffected should they choose not to participate or to withdraw during the study period.

Inclusion/exclusion: All patients will be assessed using our well established systematic evaluation protocol. Refractory asthma will be based on the definition of the American Thoracic Society Consensus Workshop. Patients recruited will have refractory asthma, will be identified as having depression using two validated questionnaires and will agree to take part and to take anti-depressant medication. Patients with poor adherence to medication, other respiratory conditions and who have had anti-depressant medication in previous the 6 months will be excluded.

Consent: People who are unable to give informed consent will be excluded from the study as they may be particularly vulnerable. Capacity to give informed consent will be assessed by the participant's usual healthcare professionals.

Risks, burdens and benefits

There is a small risk of agitation and suicidal ideation associated with commencement of selective serotonin reuptake inhibition (SSRI) anti-depressants. The investigators will attempt to minimise this risk by:

1. Contacting participants 1 week after commencing treatment and 1 week after any subsequent dose increase to ensure there is no suggestion of agitation or suicidal ideation. This is in accordance with the guidelines for initiation of SSRI therapy in adults.
2. Participants will also be contacted weekly for 2 weeks after discontinuation of study treatment. If depressive symptoms worsen patients will be advised to liaise with their GP to consider institution of treatment on clinical grounds.

ELIGIBILITY:
Inclusion Criteria:

All patients will be assessed using our well established systematic evaluation protocol. Refractory asthma will be based on the definition of the American Thoracic Society Consensus Workshop, but for the purposes of this study will be defined as follows:

* Persisting symptoms due to asthma (ACS ≥3) despite detailed assessment and management (non-adherence, alternative diagnoses and co-morbidities etc);
* Minimal maintenance therapy of high dose inhaled steroids ( ≥800 mg BDP or equivalent) long acting Beta2-agonist and / or other maintenance therapies (theophylline / leukotriene receptor antagonist).
* The requirement for maintenance oral steroids for ≥ 50% of the year or at least 3 courses of systemic steroids in the preceding 12 months.

Inclusion criteria:

* Age 18-65 years
* Refractory asthma
* Agreement to take part in trial and to take anti-depressant medication
* Hospital Anxiety and Depression Score ≥11
* Hamilton Depression Rating Scale ≥ 17

Exclusion Criteria:

* Poor adherence with medication (prescription records, ≤50% of inhaled combination filled in previous 6 months)
* Significant co-morbidity due to conditions other than asthma
* Anti-depressant medication in previous 3 months
* Pregnancy
* Patients requiring non-steroidal anti-inflammatory drugs, aspirin or warfarin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in Asthma Control Score | 12 weeks
Improvement in Hamilton Rating Scale for Depression (HDRS) | 12 weeks

SECONDARY OUTCOMES:
Improvement in Asthma Quality of Life Questionnaire (AQLQ) | 12 weeks
Improvement in Hospital Anxiety and Depression Scale (HADS) | 12 weeks
Improvement in Lung function | 12 weeks
Reduction in Fractional exhaled nitric oxide | 12 weeks
Sputum eosinophil count | 12 weeks
Reduction in dose of oral steroids (if applicable) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Respiratory Centre, Belfast City Hospital, Belfast, United Kingdom